CLINICAL TRIAL: NCT05647460
Title: Precision of Computer Guided Screw Holes Locating Guide and Custom-made Plates vs Conventional Plate Osteosynthesis in Management of Parasymphseal Mandibular Fracture
Brief Title: Computer Guided Screw Holes Locating Guide and Custom-made Plates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed abd ellati tag eldin ahmed, master degree researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3922
Record Dates: First submitted 2022-12-05; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-09

CONDITIONS: Mandibular Fractures
Keywords: parasymphseal mandibular fractures
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer guided plates (Active Comparator): computer guided screw holes locating guide and custom-made plates in management of parasymphseal mandibular fracture
  Interventions: Procedure: computer guided screw holes locating guide and custom-made plates
- conventional plates (Active Comparator): conventional plate osteosynthesis in management of parasymphseal mandibular fracture
  Interventions: Procedure: conventional plates

INTERVENTIONS:
Procedure: computer guided screw holes locating guide and custom-made plates — Virtual planning and guide fabrication for the study group:
  * Preoperative CT.
  * Virtual reduction of broken segments on software.
  * Gain occlusion.
  * Design surgical screw holes locating guide.
  * Design the custom-made plates.
  * Print the screw holes locating guide and the custom-made plate.
  * Surgical guiding tools: screw holes locating guide and custom-made plates.
  Put the specific screw holes locating device in place and drill the screw holes, remove the screw holes locating device and mobilize the segments then apply the custom-made plates and fix it with screw for passive reduction of the segments. Then suture the mentalis muscle then the mucosa.
  Arms: computer guided plates
Procedure: conventional plates — mobilize the broken segment first, Arch bar was made to achieve proper occlusion put the compression plate on the inferior border and remove it for further bending using plate pliers for further accommodation of the plate on the inferior border the fix it in place using compression and tension plate.
  Arms: conventional plates

SUMMARY:
* Preoperative CT.
* Virtual reduction of broken segments on software.
* Gain occlusion.
* Design surgical screw holes locating guide.
* Design the custom-made plates.
* Print the screw holes locating guide and the custom-made plate. under general anesthesia the parasymphseal fracture will be reduced using screw holes locating guide and the custom-made plates.

DETAILED DESCRIPTION:
Interventions 26 patients involved in this study will be divided in to two different groups, first group will be reduced using patient computer guided specific screw holes locating guide and custom-made plates.

Second group fractures will be reduced by conventional work flow.

Clinical evaluation:

A through medical and dental history followed by clinical examination was carried out for all patients. Clinical measurements were taken to ensure patient adherence to our initial inclusion criteria prior to further investigations.

A preoperative digital panoramic radiograph with 1:1 magnification was taken for each patient as a primary survey in order to exclude the presence of any lesion at the area of interest nor segment loss followed by A pre-operative CT.

Virtual planning and guide fabrication for the study group:

* Preoperative CT.
* Virtual reduction of broken segments on software.
* Gain occlusion.
* Design surgical screw holes locating guide.
* Design the custom-made plates.
* Print the screw holes locating guide and the custom-made plate.
* Surgical guiding tools: screw holes locating guide and custom-made plates.

Intra operative procedures for both groups:

• In both group: the operation will under general anesthesia with nasal intubation and oral pack, Injection of 20 cc saline adrenaline 1:00000 to 0 in the sulcus for hemostasis, Vestibular mucosal incision followed by mentalis incision in 2 planes and ensure enough cough for latter muscle suturing, Reflect the flap to visualize the broken segments.

In first group:

Put the specific screw holes locating device in place and drill the screw holes, remove the screw holes locating device and mobilize the segments then apply the custom-made plates and fix it with screw for passive reduction of the segments. Then suture the mentalis muscle then the mucosa.

In second group:

mobilize the broken segment first, Arch bar was made to achieve proper occlusion put the compression plate on the inferior border and remove it for further bending using plate pliers for further accommodation of the plate on the inferior border the fix it in place using compression and tension plate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with parasymphseal mandibular class fracture needs open reduction and internal fixation.
* Patients with medical history that did not hinder plate placement (uncontrolled diabetes) and adequate proper oral hygiene.
* Both genders males and females will be included.

Exclusion Criteria:

* • • General contraindications to surgery.

  * Patients with fresh fractures (mobile segments).
  * Patients with unfavourable nor comminuted fractures.
  * Subjected to irradiation in the head and neck area less than 1 year before fixation.
  * Untreated periodontitis.
  * Poor oral hygiene and motivation.
  * Uncontrolled diabetes.
  * Pregnant or nursing.
  * Substance abuse.
  * Psychiatric problems or unrealistic expectations.
  * Severe bruxism or clenching.
  * Immunosuppressed or immunocompromised.
  * Treated or under treatment with intravenous amino-bisphosphonates.
  * Patients participating in other studies, if the present protocol could not be properly followed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
computer tomoghraphy | 3 months .
  the Computer Tomography Will calculate the segments deviation in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed omara, Study Director — Cairo University; mona el hadidy, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- See also: Description Reginald H.B. Goodday/Management of Fractures of the Mandibular Body and Symphysis. Oral Maxillofacial Surg Clin North Am. 2013 Nov;25 — http://pubmed.ncbi.nlm.nih.gov/24021623/
- See also: Evaluation of the Accuracy of Computer-Guided Mandibular Fracture Reduction. 2015 Jul;26(5):1587-91.doi: 10.1097/ SCS.0000000000001773. — http://pubmed.ncbi.nlm.nih.gov/26163841/.
- See also: Parul Sinha , Gary Skolnick , Kamlesh B Patel , Gregory H Branham , John J Chi /A 3-Dimensional-Printed Short-Segment Template Prototype for Mandibular Fracture Repair. 2018 Sep 1;20(5):373-380 — http://pubmed.ncbi.nlm.nih.gov/29710318/
- See also: Description Scott Lovald , Bret Baack, Curtis Gaball, Garth Olson, Anna 31 Hoard/Biomechanical optimization of bone plates used in rigid fixation of mandibular symphysis fractures. 2010 Aug — http://pubmed.ncbi.nlm.nih.gov/20537782/